CLINICAL TRIAL: NCT06431464
Title: In Vivo Analysis of Tattoo Particles After Picosecond Laser Compared to Nanosecond Laser
Brief Title: Tattoo Particles: Picosecond Laser Versus Nanosecond Laser
Status: Recruiting | Type: Observational
Sponsor: Universitätsklinikum Hamburg-Eppendorf (Other)
Responsible Party: Principal Investigator, Lynhda Nguyen, Principle investigator, Universitätsklinikum Hamburg-Eppendorf
Other Study IDs: 02-24
Record Dates: First submitted 2024-02-19; First posted 2024-05-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Tattoo; Pigmentation
MeSH Terms: interventions — Weights and Measures

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Nanosecond laser: Patients with unwanted tattoos who plan a nanosecond laser treatment will be recruited for measurements using a multiphoton-tomography system.
  Interventions: Other: nanosecond laser treatment + measurement with a multiphoton tomography system
- Picosecond laser: Patients with unwanted tattoos who plan a picosecond laser treatment will be recruited for measurements using a multiphoton-tomography system.
  Interventions: Other: picosecond laser treatment + measurement with a multiphoton tomography system

INTERVENTIONS:
Other: picosecond laser treatment + measurement with a multiphoton tomography system — Patients with unwanted tattoos who plan a laser treatment will be recruited for measurements using a multiphoton-tomography system. These are scheduled 6 weeks and 12 weeks post-treatment.
  Groups: Picosecond laser
Other: nanosecond laser treatment + measurement with a multiphoton tomography system — Patients with unwanted tattoos who plan a laser treatment will be recruited for measurements using a multiphoton-tomography system. These are scheduled 6 weeks and 12 weeks post-treatment.
  Groups: Nanosecond laser

SUMMARY:
- For treating unwanted tattoos, the gold standard treatment is a nanosecond or picosecond laser. However, comparative microscopic analysis is limited. Therefore, the aim of the present study is to analysis morphological changes of tattoo particles and surrounding tissue in human skin.

ELIGIBILITY:
Inclusion Criteria:

- healthy patients who plan a laser treatment of their unwanted tattoo/ tattoos at our department

Exclusion Criteria:

* laser pretreatment of their tattoos to be treated
* pregnancy, breast feeding
* open wound on the area to be treated

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: - healthy patients who plan a laser treatment of their unwanted tattoo/ tattoos at our department
Sampling Method: Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-02-01 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
Size of intercellular spaces | 6 weeks and 12 weeks post-treatment
  Size of intercellular spaces after picosecond or nanosecond laser treatment.
Size of keratinocytes | 6 weeks and 12 weeks post-treatment
  Size of keratinocytes after picosecond or nanosecond laser treatment.
Size of tattoo particles | 6 weeks and 12 weeks post-treatment
  Size of tattoo particles after picosecond or nanosecond laser treatment.
Distribution of tattoo particles | 6 weeks and 12 weeks post-treatment
  Distribution though the epidermal and dermal layers after picosecond or nanosecond laser treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Hamburg-Eppendorf, Hamburg, Germany

REFERENCES:
- [Background] Nguyen L, Mess C, Schneider SW, Huck V, Herberger K. In vivo visualisation of tattoo particles using multiphoton tomography and fluorescence lifetime imaging. Exp Dermatol. 2022 Nov;31(11):1712-1719. doi: 10.1111/exd.14646. Epub 2022 Jul 25. PMID 35837813
- [Derived] Nguyen L, Mess C, Huck V, Schneider SW, Herberger K. Intravital Visualization of Tattoo Particles After Picosecond Laser Treatment. Skin Res Technol. 2025 Oct;31(10):e70283. doi: 10.1111/srt.70283. PMID 41137607